CLINICAL TRIAL: NCT06616714
Title: Faesiblity and Safety of Endoscopic sLeeve gastrOplasty in Patients With obEsity and inflammatoRy Bowel Disease
Brief Title: Faesiblity and Safety of Endoscopic sLeeve gastrOplasty in Patients With obEsity and nflammatoRy Bowel Disease
Acronym: FLOWER
Status: Recruiting | Type: Observational
Sponsor: Laterza Lucrezia (Other)
Responsible Party: Sponsor-Investigator, Laterza Lucrezia, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Other Study IDs: 6359
Record Dates: First submitted 2024-02-16; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Diseases; Obesity
MeSH Terms: conditions — Inflammatory Bowel Diseases; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observtional Study — Observtional Study

SUMMARY:
Obesity is classified as a body mass index (BMI) above 30 kg/m2 by the World Health Organization. Both overweight (BMI > 25 kg/m2) and obesity (BMI >30 kg/m2) have increased worldwide during the last decades: 1.46 billion of the adult population were estimated to be overweight in 2008, particularly 205 million men and 297 millions of women were estimated to be obese. Obesity is associated with lower quality of life and is linked to serious comorbidities such as type 2 diabetes mellitus, hypertension, cardiovascular diseases and several cancers. Furthermore, obesity is significantly linked to a higher mortality risk compared to normal weight individuals.

Obesity is also significantly increasing in patients with IBD. Obesity enhances the inflammatory activity in IBD, leads to longer hospitalization, and increases the possibility to develop extra intestinal manifestations. Also, the frequency of having extended systemic steroid treatment and use of antibiotics seems greater in IBD patients with obesity.

Hence, treatment and prevention of obesity, especially in IBD patients, should have high priority.

DETAILED DESCRIPTION:
This is a single center, observational, prospective clinical study. ESG is a procedure commonly performed in our center thus only patients who have indication to ESG for clinical reasons will be included and ESG will be performed as per clinical practice. Follow-up of the enrolled patients will be planned according to the routine follow-up for patients with IBD regarding timing and laboratory procedures.

All participants will undergo a lifestyle modification treatment, nutritional and psychological support as per clinical standard of practice. Investigators and study personnel from the study site will ensure that equal instructions for diet, physical activity, laboratory analysis and other procedures will be used for each patient. All patients will also perform ESG within 90 days after the enrollment and they will be followed-up for 12 months after ESG. Patients will be evaluated before, immediately after and at 1, 3, 6 and 12 months after ESG.

The total duration of this study will be about 27 months. It will take place at Fondazione Policlinico Universitario A. Gemelli IRCCS, CEMAD unit and Digestive Endoscopy unit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* BMI between 30 to 40 kg/m2
* Willingness to participate in the study and ability to comply and understand the study protocol
* Patients with steroid-free clinical remission of IBD for at least 6 months before screening as defined by HBI ≤4 for patients with Crohn's disease OR by partial Mayo score (3-point Mayo score) ≤1 with rectal bleeding subscore =0 for patients with ulcerative colitis AND no use of systemic steroids during the 6 months before screening
* Patients with a previous diagnosis of Crohn's disease or Ulcerative colitis at least 3 months before screening
* Patients with stable maintenance therapy for IBD, meaning a stable dose of mesalamine, immunosuppressants of biological drugs for at least 8 weeks before ESG (baseline).

Exclusion Criteria:

* Active Helicobacter pylori infection, causing erosions or ulcers of the stomach or duodenum.
* Organic or motility disorder of the stomach and / or esophagus
* Previous bariatric surgery or any other type of surgery that causes alteration of the lumen of the esophagus, stomach and duodenum
* Ongoing or active malignancy during the last 5 years.
* Myocardial infarction during the past 6 months or/and heart failure class III or IV according to the New York Heart association's classification.
* Drug or alcohol abuse
* Bulimic or binge eating pattern
* Uncontrolled thyroid disease
* Pregnancy, breastfeeding
* Psychiatric or cooperative problems or low compliance that is a contraindication from participating in the study.
* Liver cirrhosis of any Child-Pugh stage or MELD> 15 Chronic Severe Renal Insufficiency (eGFR < 30 ml/min/1.73 m2 based on CKD-EPI equation)
* Currently participating in other study, or previously participated in an experimental drugs trial within 30 days before or 5 half-life of the drug administered
* Active IBD as defined by HBI >4 for patients with Crohn's disease OR by partial Mayo score >1 with rectal bleeding subscore ≥1 for patients with ulcerative colitis OR by the concomitant use of systemic steroids to control disease activity in both Crohn's disease and ulcerative colitis
* Any health issue that might put the patient at risk if the treatment is performed, judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IBD in remission and obesity
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility Assessment Based on Completion Rate of ESG Procedure Without Complications | 24 month
  Feasibility will be expressed as the percentage of patients who will complete the ESG procedure without intra-procedural and post-procedural (within 48 hours) complications.

CONTACTS AND LOCATIONS:
Overall Officials: Lucrezia Laterza, PI, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS, Rome
Locations (1):
- Lucrezia Laterza, Roma, Italy